CLINICAL TRIAL: NCT05343637
Title: A Phase 2a, Dose Escalation Study to Evaluate the Effect of RT234 on Cardiopulmonary Hemodynamics in Subjects With Pulmonary Arterial Hypertension
Brief Title: A Dose Escalation Study to Evaluate the Effect of RT234 in Subjects With Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Respira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT234-CL201; ACTRN12619001178134 (Registry Identifier: Australian New Zealand Clinical Trials Registry (ANZCTR))
Record Dates: First submitted 2022-04-04; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension; Vascular Diseases; Cardiovascular Diseases; Hypertension, Pulmonary; Lung Diseases; Respiratory Tract Diseases; Vardenafil Dihydrochloride; Vasodilator Agents; Phosphodiesterase 5 Inhibitors; Phosphodiesterase Inhibitors; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension; Vascular Diseases; Cardiovascular Diseases; Hypertension, Pulmonary; Lung Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- RT234 - Cohort 1 (Experimental): Participants will receive RT234 as 0.2 mg and 0.6 mg
  Interventions: Combination Product: Drug: RT234 - vardenafil inhalation powder; Device: RS01 dry powder inhaler (RS01 DPI)
- RT234 - Cohort 2 (Experimental): Participants will receive RT234 as 0.6 mg and 1.2 mg
  Interventions: Combination Product: Drug: RT234 - vardenafil inhalation powder; Device: RS01 dry powder inhaler (RS01 DPI)
- RT234 - Cohort 3 (Experimental): Participants will receive RT234 as 1.2 mg and 2.4 mg
  Interventions: Combination Product: Drug: RT234 - vardenafil inhalation powder; Device: RS01 dry powder inhaler (RS01 DPI)

INTERVENTIONS:
Combination Product: Drug: RT234 - vardenafil inhalation powder; Device: RS01 dry powder inhaler (RS01 DPI) — RT234 is a drug/device combination product composed of vardenafil hydrochloride as the drug constituent and will utilize RS01 DPI device.
  Other Names: vardenafil inhalation powder; inhaled vardenafil

SUMMARY:
This multicenter, open label, Phase 2a study is designed to evaluate the effect of inhaled RT234 delivered in a dose escalation manner on the change in pulmonary vascular resistance (PVR) in subjects with Pulmonary Arterial Hypertension (PAH) undergoing Right heart catheterization (RHC).

This study is also known as Vardenafil Inhaled for Pulmonary Arterial Hypertension PRN Phase 2a (VIPAH-PRN 2a) study

DETAILED DESCRIPTION:
The drawbacks of current therapies and the lack of an approved as needed (PRN) treatment for PAH that improves exercise ability and quality of life, form the basis for development of RT234 (inhaled vardenafil). The current study will identify the effective dose(s) of RT234 to acutely improve pulmonary vascular hemodynamics when delivered in a dose escalation manner in subjects with World Health Organization (WHO) Group 1 PAH undergoing RHC. In addition, this study will also provide valuable efficacy and safety insights into the interactions between RT234 and background disease-specific PAH therapy on pulmonary hemodynamics and right heart function.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 80 years of age, inclusive.
2. Diagnosis of RHC-confirmed WHO Group 1 PAH in any of the following three categories: Idiopathic, primary or familial pulmonary arterial hypertension (IPAH, PPH, or FPAH); OR PAH associated with one of the following connective tissue diseases (CTD):

   1. Systemic sclerosis (scleroderma)
   2. Limited scleroderma
   3. Mixed connective tissue disease
   4. Systemic lupus erythematosus
   5. Overlap syndrome
   6. Other autoimmune disorders;

   OR PAH associated with:
   1. Human immunodeficiency virus (HIV) infection with no evidence of opportunistic infection in the preceding 6 months;
   2. Simple, congenital systemic-to-pulmonary shunts at least one-year post-surgical repair.
   3. Exposure to legal drugs, chemicals and toxins, such as fenfluramine, derivatives, other anorexigens, toxic rapeseed oil or L-tryptophan. Subjects with PAH associated with illegal drug use, such as methamphetamine, were excluded.
3. Previous diagnosis with PAH with the following conditions:

   1. Stable PAH without significant adjustments of disease-specific background PAH therapy, at least 3 months prior to RHC procedure;
   2. If on corticosteroids, has been receiving a stable dose of ≤ 20 mg/day of prednisone (or equivalent dose of other corticosteroid) for at least 30 days prior to RHC procedure.
4. Pulmonary Function Tests within 24 months prior to RHC procedure that fulfilled the following criteria (pulmonary function; (PFT may be assessed at Screening if historical PFT results are not available):

   1. Forced Expiratory volume in one second (FEV1) ≥ 60% predicted (pre-bronchodilators);
   2. FEV1/ forced expiratory vital capacity (FVC) ≥ 60% (pre-bronchodilators);
   3. FVC ≥ 60% predicted.

Exclusion Criteria:

1. Baseline systemic hypotension, defined as MAP < 50 mmHg or systolic blood pressure (SBP)< 90 mmHg at Screening.
2. Requirement of intravenous inotropes within 30 days prior to RHC procedure.
3. Use of oral, topical or inhaled nitrates within 14 days prior to RHC procedure.
4. Uncontrolled systemic hypertension: SBP > 160 mmHg or diastolic blood pressure (DBP) >100 mmHg at Screening.
5. History of portal hypertension or chronic liver disease, including active viral replication of hepatitis B and/or hepatitis C or classified as having moderate to severe hepatic impairment (Child-Pugh Class B-C).
6. Chronic renal insufficiency as defined by serum creatinine > 2.5 mg/dL at Screening or requires dialysis.
7. History of atrial septostomy.
8. Unrepaired congenital heart disease (CHD).
9. Pericardial constriction; restrictive or congestive cardiomyopathy.
10. History of left ventricular ejection fraction (EF) < 40% by multiple gated acquisition scan (MUGA), angiography, echocardiography, or cardiac magnetic resonance imaging (CMRI).
11. Symptomatic coronary disease with demonstrable ischemia.
12. Poorly controlled asthma defined by active wheezing and/or cough at the time of Screening or day of participation in Parts A and B.
13. Clinically significant intercurrent illness (including lower respiratory tract infection) or clinically significant surgery within 30 days prior to study drug administration.
14. Clinical RHC < 14 days prior to Screening.
15. History of non-arteritic anterior ischemic optic neuropathy (NAION) or retinitis pigmentosa.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of adverse events (AEs) | Screening to Day 30
  Evaluation of AEs will be measured by clinical examination and participant self-reporting. Known or possible adverse events include headache, lightheadedness and cough.
Peak plasma concentration (Cmax) | At baseline, 5, 15, 30, 45 and 60 minutes post-end of inhalation for the first RT234 dose and at 5, 15, 30, 45, 60, 75, 90, 105 and 120 minutes post-end of inhalation for the second RT234 dose.
  Change in Cmax at each dose level on Day 1.
Time to peak plasma concentration (Tmax) | At baseline, 5, 15, 30, 45 and 60 minutes post-end of inhalation for the first RT234 dose and at 5, 15, 30, 45, 60, 75, 90, 105 and 120 minutes post-end of inhalation for the second RT234 dose.
  Change in Tmax at each dose level on Day 1.
Area under the plasma concentration versus time curve (AUC) | At baseline, 5, 15, 30, 45 and 60 minutes post-end of inhalation for the first RT234 dose and at 5, 15, 30, 45, 60, 75, 90, 105 and 120 minutes post-end of inhalation for the second RT234 dose.
  Change in AUC at each dose level on Day 1.
Terminal half-life | At baseline, 5, 15, 30, 45 and 60 minutes post-end of inhalation for the first RT234 dose and at 5, 15, 30, 45, 60, 75, 90, 105 and 120 minutes post-end of inhalation for the second RT234 dose.
  Change in terminal half-life at each dose level on Day 1.
Change in pulmonary vascular resistance (PVR) | At baseline, 5, 15, 30, 45 and 60 minutes post-end of inhalation for the first RT234 dose and at 5, 15, 30, 45, 60, 75, 90, 105 and 120 minutes post-end of inhalation for the second RT234 dose on Day 1.
  Maximal change from baseline in PVR assessed at the time by right heart catheterisation (RHC).

CONTACTS AND LOCATIONS:
Overall Officials: Carol Ann Satler, MD, PhD, Study Director — Respira Therapeutics
Locations (3):
- Australia (3):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Royal Hobart Hospital, Hobart, Tasmania
  - The Alfred Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No